CLINICAL TRIAL: NCT05915000
Title: Alterations of CSF Protein Markers As Prognostic Indicator of the Response to Cerebrospinal Fluid Shunting in Chronic Hydrocephalus in Adults
Brief Title: CSF Protein Markers As Prognostic Indicators of the Response to CSF Shunt in Normotensive Hydrocephalus
Status: Recruiting | Type: Observational
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Vicente Vanaclocha, Professor, University of Valencia
Other Study IDs: 20/2023
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-06

CONDITIONS: Beta-amiloid and Phospho-tau Proteins in CSF; Ventricular Size After CSF Shunt; Cognitive Impairment and CSF Shunt; Motor Impairment Evolution After CSF Shunt
Keywords: Hydrocephalus; Normal pressure hydrocephalus; CSF shunt; Cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction; Hydrocephalus; Hydrocephalus, Normal Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Lumbar CSF protein marker determination — The cerebrospinal fluid levels of the Aβ1-42 amyloid, h-tau and phospho-tau proteins will be assessed. The response of patients to the possible implantation of a ventricular peritoneal shunt will be assessed through neuropsychological, gait and ventricular size studies assessed through cerebral magnetic resonance studies.

SUMMARY:
In all published series of adult chronic hydrocephalus, there is a percentage between twenty and twenty-five percent of patients who present poor results after implantation of a cerebrospinal fluid shunt,1-11 usually ventriculoperitoneal. The lumboperitoneal shunt is also used but much more rarely.

The diagnosis of this pathology is based on the clinical picture, neuroimaging studies (Evans index and corpus callosum angle), cerebrospinal fluid dynamics tests (Katzman test), and invasive intracranial pressure measurements. Despite all this diagnostic arsenal, there is a high percentage of patients (mentioned above) in which treatment by diversion of cerebrospinal fluid does not offer the expected results. Traditionally, this has been attributed to chronic adult hydrocephalus being associated with other types of dementia. This may be the case in some patients, and it would be important to predict which patients will not improve or who will improve poorly in the case of insertion of a cerebrospinal fluid shunt.

DETAILED DESCRIPTION:
Adult chronic hydrocephalus, also known as normal pressure hydrocephalus or normal pressure hydrocephalus, presents with the classic Hakim-Adams triad, gait ataxia or "magnetic gait", urinary incontinence, and dementia.

Most cases have an idiopathic origin and constitute the only potentially reversible cause of dementia with surgical treatment (using a system for shunting the cerebrospinal fluid or CSF from the lateral ventricles or the thecal sac to the peritoneal cavity or right atrium ), so it is especially important to diagnose and treat it properly.

The prevalence of this pathology is increasing in line with the increase in the life expectancy of the population.

The diagnosis of this pathology is based on the clinical features, neuroimaging studies (CT and Magnetic Resonance), cerebrospinal fluid dynamics tests (Katzman test), cerebrospinal fluid drainage by lumbar puncture or using lumbar drainage for hours, and invasive measurements of Intracranial Pressure (ICP). Continuous monitoring of Intracranial Pressure with the patient admitted for 3-5 days (continuously night and day) is the most sensitive and specific diagnostic method for this disease, but it also has its false positives and negatives. Likewise, even though complications are very infrequent, it is an invasive technique that requires prolonged and continuous recordings to assess hydrodynamic changes.

Unfortunately, and despite all the diagnostic arsenal, the results of treatment using cerebrospinal fluid shunts (lumboperitoneal or ventriculoperitoneal), even in the best series, yield 20-25% poor results. These poor results have been attributed to many factors, including associated cerebral vascular disease problems, coexisting dementia not always well diagnosed, and Parkinson's disease.

On the other hand, the incorrect indication of a shunt can lead to unnecessary complications, potential morbidity and mortality (subdural hematomas, infections, etc.), and the low success rates mentioned above. Therefore, it is necessary to optimize the diagnosis and treatment of these patients as much as possible.

In an attempt to improve the diagnostic arsenal and, above all, try to predict which patients will improve and in which areas (cognitive, motor, or sphincter control), some researchers have studied the levels of certain proteins or peptides. in the cerebrospinal fluid obtained by a lumbar or ventricular puncture to try to find some kind of correlation between the levels of these protein markers and the type of dementia (Alzheimer's, for example, or adult chronic hydrocephalus) and the response to be expected with the implantation of a cerebrospinal fluid shunt. The markers have been highly varied (amyloid β1-42, amyloid β1-40, T-tau, phospho-tau, neurofilament light chain protein, neurogranin, monocyte chemoattractant protein), and not all of them are available to all hospitals. In our environment, we have the determination in cerebrospinal fluid of the Aβ1-42 amyloid, phospho-tau, and h-tau proteins, which are the most widely used internationally. The purpose of this study is to try to see if there is a correlation between the levels of cerebrospinal fluid obtained by lumbar puncture during the practice of the Katzman test and the results of the implantation of a cerebrospinal fluid shunt and to try to find out which marker is related to which the improvement of each of the three symptoms that afflict patients with adult chronic hydrocephalus, that is, cognitive impairment, gait problems, and inadequate sphincter control.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years, there is no maximum age, especially if it is understood that this pathology is more frequent as one advance in age, especially among males; pathology compatible with chronic adult hydrocephalus

Exclusion Criteria:

* All patients whose suspected diagnosis is not adult chronic hydrocephalus will be excluded, specifically those with cerebrovascular disease, dementia not due to adult chronic hydrocephalus, Alzheimer's disease, Parkinson's disease, and hereditary degenerative brain pathology. Huntington's chorea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study sample will be made up only of patients who meet the suspected diagnosis of adult chronic hydrocephalus, who are the ones who are going to have the valve implanted and followed up over time. In addition, the sample will be extracted with the biomarkers. The presence or absence of these biomarkers and their levels will be correlated with the clinical evolution of the patients so that these biomarkers could be used as prognostic indicators or to early identify those subjects in whom the cause of the symptoms was not really hydrocephalus but incipient dementia of another type (or other pathology).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-06-13 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between lumbar CSF protein markers and response to CSF shunt in normal pressure hydrocephalus | 1 year
  To try to establish the positive correlation between the abnormal levels in cerebrospinal fluid of the proteins beta 1-42 amyloid, h-tau and phospho-tau and the clinical outcome before the implantation of a cerebrospinal fluid shunt system.
Lumbar CSF protein marker levels that recommend no CSF shunt in normal pressure hydrocephalus | 1 year
  If there is a positive correlation, determine which would be the abnormal levels in the cerebrospinal fluid of the proteins β1-42 amyloid, h-tau and phospho-tau in the event of which a cerebrospinal fluid shunt system should not be implanted

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital General Universitario de Valencia, Valencia, Valencia
  - Vicente Vanaclocha, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No
Publish data once the study is finished

REFERENCES:
- [Background] Braun M, Bjurnemark C, Seo W, Freyhult E, Nyholm D, Niemela V, Blennow K, Zetterberg H, Fallmar D, Kultima K, Virhammar J. Higher levels of neurofilament light chain and total tau in CSF are associated with negative outcome after shunt surgery in patients with normal pressure hydrocephalus. Fluids Barriers CNS. 2022 Feb 14;19(1):15. doi: 10.1186/s12987-022-00306-2. PMID 35164790
- [Background] Thavarajasingam SG, El-Khatib M, Vemulapalli KV, Iradukunda HAS, Laleye J, Russo S, Eichhorn C, Eide PK. Cerebrospinal fluid and venous biomarkers of shunt-responsive idiopathic normal pressure hydrocephalus: a systematic review and meta-analysis. Acta Neurochir (Wien). 2022 Jul;164(7):1719-1746. doi: 10.1007/s00701-022-05154-5. Epub 2022 Mar 1. PMID 35230552
- [Background] Said HM, Kaya D, Yavuz I, Dost FS, Altun ZS, Isik AT. A Comparison of Cerebrospinal Fluid Beta-Amyloid and Tau in Idiopathic Normal Pressure Hydrocephalus and Neurodegenerative Dementias. Clin Interv Aging. 2022 Apr 11;17:467-477. doi: 10.2147/CIA.S360736. eCollection 2022. PMID 35431542
- [Background] Pyrgelis ES, Boufidou F, Constantinides VC, Papaioannou M, Papageorgiou SG, Stefanis L, Paraskevas GP, Kapaki E. Cerebrospinal Fluid Biomarkers in iNPH: A Narrative Review. Diagnostics (Basel). 2022 Nov 28;12(12):2976. doi: 10.3390/diagnostics12122976. PMID 36552981
- [Background] Darrow JA, Lewis A, Gulyani S, Khingelova K, Rao A, Wang J, Zhang Y, Luciano M, Yasar S, Moghekar A. CSF Biomarkers Predict Gait Outcomes in Idiopathic Normal Pressure Hydrocephalus. Neurol Clin Pract. 2022 Apr;12(2):91-101. doi: 10.1212/CPJ.0000000000001156. PMID 35733946
- [Background] Lukkarinen H, Tesseur I, Pemberton D, Van Der Ark P, Timmers M, Slemmon R, Janssens L, Streffer J, Van Nueten L, Bottelbergs A, Rauramaa T, Koivisto AM, Herukka SK, Korhonen VE, Junkkari A, Hiltunen M, Engelborghs S, Blennow K, Zetterberg H, Kolb HC, Leinonen V. Time Trends of Cerebrospinal Fluid Biomarkers of Neurodegeneration in Idiopathic Normal Pressure Hydrocephalus. J Alzheimers Dis. 2021;80(4):1629-1642. doi: 10.3233/JAD-201361. PMID 33720890
- [Background] Kawamura K, Miyajima M, Nakajima M, Kanai M, Motoi Y, Nojiri S, Akiba C, Ogino I, Xu H, Kamohara C, Yamada S, Karagiozov K, Ikeuchi T, Kondo A, Arai H. Cerebrospinal Fluid Amyloid-beta Oligomer Levels in Patients with Idiopathic Normal Pressure Hydrocephalus. J Alzheimers Dis. 2021;83(1):179-190. doi: 10.3233/JAD-210226. PMID 34275898
- [Background] Hua R, Liu C, Liu X, Zhu J, Zhang J, Wang L, Shi Z, Li J, Kong S, Yang C, Liu N, Liu L, Sun J, Yang Q, Wu Y, Zhou Y, Li Y, Xing Y. Predictive Value of Cerebrospinal Fluid Biomarkers for Tap Test Responsiveness in Patients With Suspected Idiopathic Normal Pressure Hydrocephalus. Front Aging Neurosci. 2021 May 20;13:665878. doi: 10.3389/fnagi.2021.665878. eCollection 2021. PMID 34093167
- [Background] Jingami N, Uemura K, Asada-Utsugi M, Kuzuya A, Yamada S, Ishikawa M, Kawahara T, Iwasaki T, Atsuchi M, Takahashi R, Kinoshita A. Two-Point Dynamic Observation of Alzheimer's Disease Cerebrospinal Fluid Biomarkers in Idiopathic Normal Pressure Hydrocephalus. J Alzheimers Dis. 2019;72(1):271-277. doi: 10.3233/JAD-190775. PMID 31561378
- [Background] Jeppsson A, Wikkelso C, Blennow K, Zetterberg H, Constantinescu R, Remes AM, Herukka SK, Rauramaa T, Nagga K, Leinonen V, Tullberg M. CSF biomarkers distinguish idiopathic normal pressure hydrocephalus from its mimics. J Neurol Neurosurg Psychiatry. 2019 Oct;90(10):1117-1123. doi: 10.1136/jnnp-2019-320826. Epub 2019 Jun 5. PMID 31167811
- [Background] Nakajima M, Miyajima M, Ogino I, Akiba C, Kawamura K, Kamohara C, Fusegi K, Harada Y, Hara T, Sugano H, Tange Y, Karagiozov K, Kasuga K, Ikeuchi T, Tokuda T, Arai H. Preoperative Phosphorylated Tau Concentration in the Cerebrospinal Fluid Can Predict Cognitive Function Three Years after Shunt Surgery in Patients with Idiopathic Normal Pressure Hydrocephalus. J Alzheimers Dis. 2018;66(1):319-331. doi: 10.3233/JAD-180557. PMID 30248058
- [Background] Akiba C, Nakajima M, Miyajima M, Ogino I, Motoi Y, Kawamura K, Adachi S, Kondo A, Sugano H, Tokuda T, Irie K, Arai H. Change of Amyloid-beta 1-42 Toxic Conformer Ratio After Cerebrospinal Fluid Diversion Predicts Long-Term Cognitive Outcome in Patients with Idiopathic Normal Pressure Hydrocephalus. J Alzheimers Dis. 2018;63(3):989-1002. doi: 10.3233/JAD-180059. PMID 29710721
- [Background] Chen Z, Liu C, Zhang J, Relkin N, Xing Y, Li Y. Cerebrospinal fluid Abeta42, t-tau, and p-tau levels in the differential diagnosis of idiopathic normal-pressure hydrocephalus: a systematic review and meta-analysis. Fluids Barriers CNS. 2017 May 10;14(1):13. doi: 10.1186/s12987-017-0062-5. PMID 28486988
- [Background] Craven CL, Baudracco I, Zetterberg H, Lunn MPT, Chapman MD, Lakdawala N, Watkins LD, Toma AK. The predictive value of T-tau and AB1-42 levels in idiopathic normal pressure hydrocephalus. Acta Neurochir (Wien). 2017 Dec;159(12):2293-2300. doi: 10.1007/s00701-017-3314-x. Epub 2017 Sep 9. PMID 28889317